CLINICAL TRIAL: NCT04337203
Title: SHARE-S Aim 3: Shared Healthcare Actions & Reflections Electronic Systems in Survivorship
Brief Title: Shared Healthcare Actions and Reflections Electronic Systems in Survivorship
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00064683; WFBCCC 99420 (Other: Wake Forest Baptist Comprehensive Cancer Center); 1P50CA244693-01 (NIH)
Record Dates: First submitted 2020-04-01; First posted 2020-04-07 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Cancer; Survivorship; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHARE-S (Experimental): Three components consisting of electronic referral, health coaching and tailored text/email messages for patients that have been referred to the cancer survivorship clinic.
  Interventions: Behavioral: SHARE-S Implementation Program

INTERVENTIONS:
Behavioral: SHARE-S Implementation Program — The program consists of three components: An electronic referral among clinical teams for potential participants, patient engagement with survivorship care planning guidelines through self-management/health coaching. One coaching call before a clinic visit (60 minutes) and two coaching calls after the clinic visit (30 minutes each). Participants will also receive automated, tailored text messages (daily for three weeks before and after a clinic visit for a total of six weeks).

SUMMARY:
The primary purpose of this study is conduct a pilot study testing the study protocols, implementation program, and mixed-methods data collection.

DETAILED DESCRIPTION:
Primary Objectives:

• To evaluate how successfully SHARE-S can be implemented into clinical care as characterized by rates of enrollment. Investigators hypothesize >30% of patients e-referred to SHARE-S will enroll.

Secondary Objectives:

* To assess additional implementation outcomes that evaluate preliminary implementation success (i.e., further assessment of adoption, acceptability, appropriateness, further assessment of feasibility, and fidelity).
* To describe service outcome variability to inform future studies. Investigators will assess service outcomes relevant to Commission on Cancer requirements by reporting annual estimates for: (1) the estimated number of patients impacted by SHARE-S; (2) the cancer sites impacted by SHARE-S; and the (3) resources/processes utilized to enhance each of the chosen services if barriers were encountered. We will also assess safety and perceived patient-centeredness of care.
* To describe patient health outcome variability to inform future studies (i.e., social role, physical functioning, anxiety, depression, fatigue, sleep disturbance, pain, cancer-specific quality of life, health behaviors, patient autonomy, self-efficacy for managing cancer, engagement with the survivorship care plan document, and satisfaction with care).
* To evaluate the Implementation Program we will assess key milestones and processes for this pilot study of the Implementation Stage measured at the clinic level.
* To qualitatively assess implementation barriers and facilitators using semi-structured interviews that will be audio-recorded.
* To examine how study results vary by cancer type.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Documented or planned cancer survivorship visit
* Have a texting enabled telephone
* Cognitively able to complete study procedures as judged by the study team
* Able to understand, read and write English

Children under the age of 18 with cancer will be excluded due to the potentially different self-management support intervention needs of this population that will likely include parental involvement. Results from this research may inform future studies in children with cancer under 18 who should be researched separately.

Exclusion Criteria

- Declined participation in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Sohl, Ph.D, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SHARE-S Intervention: SHARE-S Intervention
Period: Overall Study
Arm/Group | SHARE-S Intervention
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: Intervention
Arm/Group | Single Arm
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 29
  More than one race | 0
  Unknown or Not Reported | 1
BMI, Continuous [Mean (Standard Deviation); unit: Kg/m^2] | 32.2 (6.8)
Marital Status, Categorical [Count of Participants; unit: Participants]
  Currently Married | 28
  Separated | 1
  Divorced | 3
  Widowed | 2
  Single, never married | 5
  Prefer not to answer | 1
Highest Grade, Categorical [Count of Participants; unit: Participants]
  8th to 11th grade | 1
  High school or equivalent | 5
  Vocation/technical school post HS | 1
  Associate's degree/some college | 8
  Bachelor's degree | 17
  Graduate or professional school | 8
Primary Tumor Site, Categorical [Count of Participants; unit: Participants]
  Breast | 18
  Colorectal | 1
  Endometrial | 3
  Non-Hodgkin Lymphoma | 1
  Prostate | 10
  Other | 7
History of Cancer-Related Surgical Procedure, Categorical [Count of Participants; unit: Participants]
  Yes | 25
  No | 15
History of Radiation Therapy, Categorical [Count of Participants; unit: Participants]
  Yes | 28
  No | 12
History of Chemotherapy, Categorical [Count of Participants; unit: Participants]
  Yes | 18
  No | 22
Time since last treatment/surgery (months) [Median (Inter-Quartile Range); unit: months] | 5 [2 to 39]
Difficult to pay monthly bills, Categorical [Count of Participants; unit: Participants]
  Very difficult | 2
  Somewhat difficult | 8
  Not very difficult | 16
  Not at all difficult | 14
Travel to clinic bills (minutes) [Mean (Standard Deviation); unit: minutes] | 31.5 (28.6)
Use internet or email at least occasionally, Categorical [Count of Participants; unit: Participants]
  Yes | 38
  No | 2
Confident filling out medical forms, Categorical [Count of Participants; unit: Participants]
  Extremely | 27
  Quite a bit | 11
  Somewhat | 2
  A little bit | 0
  Not at all | 0
Number of times received income assistance, Categorical [Count of Participants; unit: Participants]
  Never | 30
  Once | 4
  Twice | 4
  Three times | 1
  Four times | 0
  More than four times | 1
Rural residence, Categorical [Count of Participants; unit: Participants]
  Yes | 5
  No | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Enrolled Out of Those Electronically Referred
Description: Using a 95% confidence interval (CI) to determine the range of estimates that are consistent with our data. Investigators will track the number of new patients seen in the Survivorship Clinic, and the percent who agree to be referred to SHARE-S.
Time Frame: 1 year, 8 months
Population: Total number reflects the total number of participants who were electronically referred in SHARE-S intervention.
Measure: Number (95% Confidence Interval); unit: number of participants
Groups:
- SHARE-S Intervention: Enrolled in intervention
Arm/Group | SHARE-S Intervention
Number analyzed (Participants) | 118
number of participants | 40 [29 to 50]
Statistical Analysis 1: Comparison: SHARE-S Intervention; Test type: Other — Feasibility study and calculated confidence interval; p = 0.54, Independent samples proportions test

2. Secondary Outcome: Adoption - Number of Electronically Referred Patients - Those Possible [Based on Chart Review]
Description: Using a 95% confidence interval to determine the range of estimates that are consistent with our data. Investigators will track the number of new patients seen in the Survivorship Clinic, and the percent who agree to enroll in SHARE-S
Time Frame: 1 year, 8 months
Population: Total number given a care plan
Measure: Count of Participants; unit: Participants
Groups:
- SHARE-S - Intervention: Participants given a care plan
Arm/Group | SHARE-S - Intervention
Number analyzed (Participants) | 409
Participants | 118

3. Secondary Outcome: Acceptability of Intervention Measure
Description: This measure will be used along with qualitative feedback among participants using a mixed-methods to assess acceptability of intervention with different cancer types. Acceptability ranges from 1-5 with higher scores indicating more acceptability.
Time Frame: Up to 30 days after the final intervention session.
Population: Initial cohort less 6 lost to follow-up at time of subsequent survey administration
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SHARE-S Intervention: Initial cohort less 6 lost to follow-up at time of subsequent survey administration
Arm/Group | SHARE-S Intervention
Number analyzed (Participants) | 34
score on a scale | 4.4 (.6)

4. Secondary Outcome: Appropriateness of Intervention Measure
Description: This measure will be used along with qualitative feedback among participants using a mixed-methods to assess appropriateness of intervention with different cancer types. Appropriateness ranges from 1-5 with higher scores meaning more appropriateness.
Time Frame: Up to 30 days after the final intervention session.
Population: Initial cohort less 6 lost to follow-up at time of subsequent survey administration
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SHARE-S Intervention
Number analyzed (Participants) | 34
score on a scale | 4.3 (0.6)

5. Secondary Outcome: Number of Participants Enrolled Per Month
Description: This will be defined as the average number of participants that enroll per month that the study is open to enrollment.
Time Frame: 1 year, 8 months
Population: Number enrolled per month.
Measure: Mean (Full Range); unit: participants/month
Groups:
- SHARE-S Intervention: SHARE-S Intervention Enrolled Participants
Arm/Group | SHARE-S Intervention
Number analyzed (Participants) | 40
participants/month | 2 [0 to 7]

6. Secondary Outcome: Feasibility of Intervention Measure
Description: This measure will be used along with qualitative feedback among participants using a mixed-methods to assess feasibility of intervention with different cancer types. Feasibility ranges from 1-5 with higher scores indicating more feasibility.
Time Frame: Up to 30 days after the final intervention session.
Population: Initial cohort less 6 lost to follow-up at time of subsequent survey administration
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SHARE-S Intervention
Number analyzed (Participants) | 34
score on a scale | 4.3 (.5)

7. Secondary Outcome: Retention Rates
Description: Retention is defined as participants that complete the follow up assessment.
Time Frame: Up to 30 days after the final intervention session.
Population: SHARE-S Intervention enrolled participants less 5 lost in follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | SHARE-S Intervention
Number analyzed (Participants) | 40
Participants | 35

8. Secondary Outcome: Number of Participants Adhering to Text Responses
Description: Defined as participants that adhere to responding to text messages received during intervention.
Time Frame: 1 year, 8 months
Population: 40 enrolled
Measure: Count of Participants; unit: Participants
Groups:
- SHARE-S Intervention: Participants enrolled in the intervention.
Arm/Group | SHARE-S Intervention
Number analyzed (Participants) | 40
Participants | 27

9. Secondary Outcome: Participant Adherence to Coaching Sessions
Description: Defined as adherence to completing coaching sessions during the intervention.
Time Frame: 1 year, 8 months
Population: 40 enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | SHARE-S Intervention
Number analyzed (Participants) | 40
Participants | 36

10. Secondary Outcome: Length of Coaching Sessions
Description: Defined as how long each completed coaching sessions lasted during the intervention.
Time Frame: Up to 30 days after the final intervention session.
Population: 40 enrolled (mean minutes over coach calls at 3 timepoints).
Measure: Mean (Full Range); unit: minutes
Arm/Group | SHARE-S Intervention
Number analyzed (Participants) | 40
minutes | 39 [7 to 69]

11. Secondary Outcome: Number of Coaching Sessions Completed
Description: Defined as an observational checklist completed for a subset of coaching sessions.
Time Frame: 1 year, 8 months
Population: 40 enrolled
Measure: Number; unit: sessions
Arm/Group | SHARE-S Intervention
Number analyzed (Participants) | 40
sessions | 111

12. Secondary Outcome: Total Number of Patients Enrolled
Description: Number of patients enrolled will be defined as overall participants for the entirety of the study.
Time Frame: 1 year, 8 months
Population: 40 participants enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | SHARE-S Intervention
Number analyzed (Participants) | 40
Participants | 40

13. Secondary Outcome: Frequency of Adverse Events
Description: Adverse events related to the intervention will be assessed in adverse event log.
Time Frame: Up to 30 days after the final intervention session.
Population: 40 participants enrolled
Measure: Number; unit: events
Arm/Group | SHARE-S Intervention
Number analyzed (Participants) | 40
events | 0

14. Secondary Outcome: HEAL Patient-Provider Connection
Description: Patient reported measure of patient-centered communication/relatedness completed only at follow-up. Range 0-35 with higher scores indicating better communication.
Time Frame: Up to 30 days after the final intervention session.
Population: Initial cohort with 6 lost to follow-up at time of subsequent survey administration
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SHARE-S Intervention: Initial cohort with 6 lost to follow-up at time of subsequent survey administration
Arm/Group | SHARE-S Intervention
Number analyzed (Participants) | 34
score on a scale | 32.3 (4.2)

15. Secondary Outcome: Patient-Reported Health Outcomes PROMIS Profile 29
Description: Questionnaire to assess the social role (0-100), physical functioning (0-100), anxiety (0-100), depression (0-100), fatigue (0-100), sleep disturbance (0-100), pain interference (0-100), pain intensity (0-10). Lower scores indicate less of construct.
Time Frame: At baseline and up to 30 days after the final intervention session.
Population: 40 enrolled at baseline; 35 available at follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SHARE-S Intervention - Baseline: Entire sample of 40 participants responses at baseline survey
- SHARE-S Intervention - Follow-Up: Same cohort with 5 lost to follow-up at time of subsequent survey administration
Arm/Group | SHARE-S Intervention - Baseline | SHARE-S Intervention - Follow-Up
Number analyzed (Participants) | 40 | 35
score on a scale
  physical function (0-100) | 48.4 (8.2) | 49.2 (8.5)
  anxiety (0-100) | 50.6 (9.8) | 49.0 (8.5)
  depression (0-100) | 48.1 (9.3) | 45.9 (7.7)
  fatigue (0-100) | 51.3 (10.9) | 49.2 (11.5)
  sleep disturbance (0-100) | 49.6 (7.4) | 48.9 (6.3)
  social roles (0-100) | 51.2 (9.4) | 54.2 (10.8)
  pain interference (0-100) | 51.5 (10.2) | 50.3 (9.3)
  pain intensity (0-10) | 2.7 (2.4) | 2.5 (2.4)

16. Secondary Outcome: 36-Item Short Form Survey (SF-36)
Description: Participants will only answer the single item question that provides an indication of perceived change in health. Score range: 1 - excellent health, 2 - very good health, 3 - good health, 4 - fair health and 5 - poor health.
Time Frame: At baseline and up to 30 days after the final intervention session.
Population: 40 enrolled at baseline; 35 answered follow-up questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SHARE-S Intervention - Baseline | SHARE-S Intervention - Follow-Up
Number analyzed (Participants) | 40 | 35
score on a scale | 3.15 (0.83) | 3.15 (0.89)

17. Secondary Outcome: Cancer-specific Quality of Life in Adult Cancer Survivors (QLACS) Questionnaire
Description: Investigators will only assess the quality of life of adult cancer survivors measuring domains of cancer survivorship that are cancer-specific. Cancer-Specific Quality of Life (range 15-105) - higher score indicates more quality of life; Benefits of Having Cancer (range 4-28) - higher score indicates more benefits; Positive Feelings (range 4-28) - lower score indicates more positive feelings.
Time Frame: At baseline and up to 30 days after the final intervention session.
Population: 40 participants at baseline; 35 participants answered follow-up questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SHARE-S Intervention - Baseline | SHARE-S Intervention - Follow-Up
Number analyzed (Participants) | 40 | 35
score on a scale
  Cancer-Specific Quality of Life | 47 (20.5) | 40.9 (19.1)
  Benefits of Having Cancer | 13.9 (5.8) | 12.2 (5.7)
  Positive Feelings | 10.6 (5.4) | 9.5 (4.3)

18. Secondary Outcome: Index of Autonomous Functioning - Self Congruence Subscale Only
Description: The Index of Autonomous Functioning - self congruence subscale only. 5 Items were paired with a Likert-type scale with 1 = "not at all true", 2 = "a bit true", 3 = "somewhat true", 4 = "mostly true", and 5 = "completely true." Mean score is average of 5 items. Higher mean score indicate a higher level of self congruence functioning.
Time Frame: At baseline and up to 30 days after the final intervention session.
Population: 40 participants at baseline; 35 participants answered follow-up questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SHARE-S Intervention - Baseline | SHARE-S Intervention - Follow-Up
Number analyzed (Participants) | 40 | 35
score on a scale | 4.3 (.5) | 4.3 (.6)

19. Secondary Outcome: Self-Efficacy to Manage Chronic Disease Questionnaire
Description: A questionnaire made up of 6-items on a visual analog scale, ranging from 1 (not at all confident) to 10 (totally confident). Higher the mean score indicates higher self-efficacy.
Time Frame: At baseline and up to 30 days after the final intervention session.
Population: 40 participants at baseline; 35 participants answered follow-up questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SHARE-S Intervention - Baseline | SHARE-S Intervention - Follow-Up
Number analyzed (Participants) | 40 | 35
score on a scale | 7.7 (1.8) | 7.8 (1.9)

20. Secondary Outcome: Engagement With the Survivorship Care Plan
Description: Self-reported use of the care plan since enrolled on the study.
Time Frame: 1 year, 8 months
Population: 34 participants available at follow-up
Measure: Count of Participants; unit: Participants
Groups:
- SHARE-S Intervention - Follow-up: Initial baseline cohort with 6 lost to follow-up at time of subsequent survey administration
Arm/Group | SHARE-S Intervention - Follow-up
Number analyzed (Participants) | 34
Participants | 34

21. Secondary Outcome: Satisfaction of Care
Description: Participants will evaluate their overall satisfaction with their care after the study intervention. Mean of Likert scale. 1=very poor, 5=very good.
Time Frame: Up to 30 days after the final intervention session.
Population: Follow-up only
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SHARE-S Intervention - Follow-Up: Initial baseline cohort with 5 lost to follow-up at time of subsequent survey administration
Arm/Group | SHARE-S Intervention - Follow-Up
Number analyzed (Participants) | 35
score on a scale | 4.8 (.4)

22. Secondary Outcome: Health Behaviors Questionnaire - Tobacco Use
Description: Participants will be asked about their tobacco use within the last seven days. Tobacco use is scored 1=yes, 0=no. Higher values represent more participants were tobacco users.
Time Frame: At baseline and up to 30 days after the final intervention session.
Population: 40 participants at baseline; 34 participants answered follow-up questionnaire
Measure: Count of Participants; unit: Participants
Groups:
- SHARE-S Intervention - Follow-Up: Same cohort with 6 lost to follow-up at time of subsequent survey administration
Arm/Group | SHARE-S Intervention - Baseline | SHARE-S Intervention - Follow-Up
Number analyzed (Participants) | 40 | 34
Participants | 1 | 1

23. Secondary Outcome: Health Behaviors Questionnaire - Alcohol Use Disorder
Description: Participants will be asked individual questions about their alcohol use. Alcohol use disorder is on a scale of 0-12 with higher scores indicating more hazardous; men ≥ 4, women ≥ 3 is considered hazardous.
Time Frame: At baseline and up to 30 days after the final intervention session.
Population: Entire cohort at baseline; 34 participants at follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SHARE-S Intervention - Baseline | SHARE-S Intervention - Follow-Up
Number analyzed (Participants) | 40 | 34
score on a scale | 1.4 (1.9) | 1.2 (1.6)

24. Secondary Outcome: Health Behaviors Questionnaire - Physical Activity
Description: Participants will be asked individual questions about their physical activity. Physical activity is minutes/week with <90 minutes considered insufficient.
Time Frame: At baseline and up to 30 days after the final intervention session.
Population: Entire cohort at baseline; 34 participants at follow-up.
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | SHARE-S Intervention - Baseline | SHARE-S Intervention - Follow-Up
Number analyzed (Participants) | 40 | 34
minutes/week | 124.5 (140) | 162.4 (157.2)

25. Secondary Outcome: Health Behaviors Questionnaire - Fruit and Vegetable Intake
Description: Participants will be asked individual questions about their fruit and vegetable intake. Mean for the responses were calculated in cups so ½ to 1 cup = 0.75 cups, at least 2-3 cups for both considered sufficient.
Time Frame: At baseline and up to 30 days after the final intervention session.
Population: Entire cohort at baseline; 34 participants at follow-up.
Measure: Mean (Standard Deviation); unit: cups/day
Arm/Group | SHARE-S Intervention - Baseline | SHARE-S Intervention - Follow-Up
Number analyzed (Participants) | 40 | 34
cups/day | 2.7 (1.2) | 3.2 (1.6)

26. Secondary Outcome: Health Behaviors Questionnaire - Mindfulness Practice
Description: Participants will be asked individual questions how many days/week they practice mindfulness.
Time Frame: At baseline and up to 30 days after the final intervention session.
Population: Entire cohort at baseline; 34 participants at follow-up.
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | SHARE-S Intervention - Baseline | SHARE-S Intervention - Follow-Up
Number analyzed (Participants) | 40 | 34
days/week | 1.8 (2.1) | 3.4 (2.1)

ADVERSE EVENTS:
Time Frame: Up to 30 days after the final intervention session.
Groups:
- Overall: Single Arm - Intervention
Arm/Group | Overall
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT04337203/Prot_SAP_001.pdf
  • Informed Consent Form (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT04337203/ICF_000.pdf